CLINICAL TRIAL: NCT02830867
Title: Review of French Cases of Glutathione Synthetase Deficiency
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6245
Record Dates: First submitted 2016-06-17; First posted 2016-07-13 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2016-01

CONDITIONS: The Glutathione Synthetase Deficiency
Keywords: glutathione; glutathione synthetase deficiency; autosomal inheritance; recessive
MeSH Terms: conditions — Glutathione synthetase deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The glutathione synthetase deficiency, inborn error of metabolism of autosomal recessive inheritance, is a rare disease (70 patients described in the world). The outcome of these patients and potential complications of this disease are not, to date, yet all known and described.

ELIGIBILITY:
Inclusion criteria:

* All patients followed in the French hospital centers the diagnosis of glutathione synthetase deficiency has been proven by assay of residual enzyme activity or identifying a mutation of the glutathione synthetase gene

Exclusion criteria:

* No formal proof of glutathione synthetase deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients followed in the French hospital centers the diagnosis of glutathione synthetase deficiency has been proven by assay of residual enzyme activity or identifying a mutation of the glutathione synthetase gene
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Immunologically determining human acid glutathione S-transferase in a human assay sample | 1 hour after hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Service D'Urgences Medicales Pediatriques, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No